CLINICAL TRIAL: NCT05893316
Title: Hematuria Evaluation by Whole-genome Sequencing of Urine-Exfoliated Cell DNA, A Prospective, Multi-center Study
Brief Title: UroCAD for Hematuria Evaluation--A Prospective, Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Tongji Hospital (Other); RenJi Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, M. D., Changhai Hospital
Other Study IDs: CH-Hematuria-CIN
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Hematuria; Urothelial Carcinoma
Keywords: non-invasive; urothelial carcinoma; hematuria evaluation
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples were collected form each patient and DNA was extracted form urine exfoliated cells for sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hematuria patients: Hematuria patients (≥ 3 RBCs/HPF) with treatment-naïve, pathology-confirmed urothelial carcinoma or benign genitourinary system disease or with undetermined lesion presented with hematuria.
  Interventions: Diagnostic Test: urine sample collection
- Non-hematuria patients: Patients without hematuria and diagnosed with pathology-confirmed cancer other than urothelial cancer.
  Interventions: Diagnostic Test: urine sample collection

INTERVENTIONS:
Diagnostic Test: urine sample collection — The level of CIN The extracted DNA from urine exfoliated cells will be analyzed by UroCAD to determine the level of CIN.

SUMMARY:
Hematuria is recognized as an important sigh of potential urinary tract malignancy. Therefore, understanding the disease processes and discovering the potential urothelial carcinoma (UC) underlying this important sign is critical. Cystoscopy, urine cytology and imaging are most reliable methods for UC diagnosis, but certain drawbacks exist for these methods, such as invasiveness or inaccuracy. Chromosomal instability (CIN) is a hallmark of human cancer, and it's related with tumor stage and grade. Previous research has proved that analyzing CIN of the DNA extracted from urothelial cells in urine samples seems a promising method for detecting UC. Here we intend to assess CIN's performance for hematuria evaluation.

DETAILED DESCRIPTION:
Hematuria is defined as the presence of 3 or more red blood cells per high-power field (RBC/HPF) under microscopic examination of the urine, which is an important sigh of genitourinary system disease, especially UC. Several methods can be adopted for hematuria evaluation. Cystoscopy is a key component of the hematuria evaluation because it is a reliable way to evaluate the bladder and urethra. Biopsy can also be performed through cystoscopy, making it the "gold standard" for bladder cancer diagnosis. Despite its high reliability and accuracy, it's an invasive examination related with complications such as injury to the urethra, infection, and discomfort. Flat lesions may also be omitted under cystoscopy. Urine cytology is another important method for UC evaluation, but it has a sensitivity of only 15.8%-54.5%.

CIN refers to the ongoing acquisition of genomic alterations, it can range from point mutations to small-scale genomic alterations and gross chromosomal rearrangements. 60%-80% of human tumors exhibit chromosomal abnormalities suggestive of CIN. CIN is presented in UC and it has been adopted as a diagnostic method for UC, such as UroVysion test. Previously, CIN detected by low-coverage whole genome sequencing proved to be a reliable method for UC diagnosis and was named as Urine Exfoliated Cells Copy Number Aberration Detector (UroCAD). In this prospective, multi-canter, observational clinical trial, we intend to assess the possibility of UroCAD as an additional diagnostic tool for hematuria patients by collecting and analyzing 30 ml of urine sample from hematuria patient across 5 centers.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years and signed informed consent form.
* Participants presented with hematuria (≥ 3 RBCs/HPF) and meet one of the following criteria:

  1. Patients recommended to undergo cystoscopy or ureteroscopy;
  2. Patients with treatment-naïve, pathology-confirmed urothelial carcinoma;
  3. Patients diagnosed with benign genitourinary disease.
* Participants diagnosed with cancer other than urothelial carcinoma.

Exclusion Criteria:

* Participants with history of urothelial carcinoma.
* Participants with urothelial carcinoma accompanied by other malignancy.
* Individuals unwilling to sign the consent form or unwilling to provide urine sample for test or quality of urine sample is poor.
* Patients unsuitable for this clinical trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presented with hematuria (≥ 3 RBCs/HPF) and patients with malignancy other than urothelial carcinoma in Changhai Hospital, Tongji Hospital, Renji Hospital, First Affiliated Hospital of Xian Jiaotong University, and Gulou Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity | through study completion, an average of 8 months
  Comparison of the sensitivity of the UroCAD analysis versus clinically-acceptable threshold, defined as 75%.
specificity | through study completion, an average of 8 months
  Comparison of the specificity of the UroCAD analysis versus clinically-acceptable threshold, defined as 95%.
Sensitivity among hematuria patients | through study completion, an average of 8 months
  Sensitivity of UroCAD in detecting urothelial carcinoma among hematuria patients
Specificity among hematuria patients | through study completion, an average of 8 months
  Specificity of UroCAD in detecting urothelial carcinoma among hematuria patients

SECONDARY OUTCOMES:
Comparison of Sensitivity | through study completion, an average of 8 months
  Comparison of the sensitivity of the UroCAD analysis versus urine cytology
Comparison of Specificity | through study completion, an average of 8 months
  Comparison of the Specificity of the UroCAD analysis versus urine cytology

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not public for privacy protection purpose. Data without private information may be provided on request.

REFERENCES:
- [Background] Sansregret L, Vanhaesebroeck B, Swanton C. Determinants and clinical implications of chromosomal instability in cancer. Nat Rev Clin Oncol. 2018 Mar;15(3):139-150. doi: 10.1038/nrclinonc.2017.198. Epub 2018 Jan 3. PMID 29297505
- [Background] McDougal, W. Scott, et al. Campbell-Walsh urology 11th Edition review e-book. Elsevier Health Sciences, 2015.